CLINICAL TRIAL: NCT05424068
Title: Project 3 - Phase II, Preference Based, Randomized Controlled Trial of Group-Based, In Person Versus Virtual, Cancer Rehabilitation for People With Metastatic / Advanced Breast or Colorectal Cancers
Brief Title: Rehabilitation for People With Advanced Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-5539
Record Dates: First submitted 2022-04-13; First posted 2022-06-21 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Advanced Breast Cancer; Advanced Colorectal Cancer; Cancer Rehabilitation
Keywords: Cancer Rehabilitation; Virtual Cancer Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard best cancer practice (No Intervention): All participants (intervention arms 1 and 2, and control) will receive usual oncology care by their health care providers which includes recommendations for general aerobic and resistance exercise. Participants in the control group will be of recommended to work towards the recommended 90 minutes moderate to vigorous aerobic exercise, and two days a week of large muscle group strength training as recommended by the ACSM. A general brochure will be provided to all control participants providing education in line with current standard of care. This safety precautions noted these will be indicated brochure will have an open text field on the back which will allow the kinesiologist to provide and general advice at each time point. If there are particular here. Participants in all study arms may also be referred by treating health care providers to usual supportive care or early palliative care services at any time deemed necessary, and will be recorded as part of monthly data collection.
- In-person Intervention arm (Experimental): The in-person intervention arm is an 8-week program and four week short maintenance period. This includes 1 hr of in-person, group-based exercise guided by a qualified exercise professional followed by 1 hr of in-person, group based, self-management education provided by a rehabilitation expert to occur immediately following the exercise session. Each participant is given a FitBit® to track steps, heart rate and sleep. Each site (i.e., Toronto and Vancouver) will run independent, in-person exercise and educational programs based on local referrals. Self management sessions include 8 high priority topics for advanced cancer patients including: 1) goal setting, 2) managing pain, 3) reducing fatigue and improving sleep, 4) boosting brain health, 5) eating and cooking for wellness, 6) managing emotions, 7) being mindful, and 8) planning for the future. Education sessions will be run by local experts at each site.
  Interventions: Behavioral: In-person rehabilitaiton group
- Virtual Intervention arm (Experimental): The virtual intervention arm will be an 8-week program plus four week short maintenance period but will include two separate 1 hour sessions per week. This includes: 1) 60 minutes of virtual, group-based, synchronous exercise over a virtual secure platform; and, 2) A separate 60 min virtual synchronous education session provided on a separate day (to prevent virtual fatigue). 3) Encouragement to participate in a home program the other days of the week, striving for the recommended 90 min of moderate to vigorous aerobic exercise and 2 days of week or resistance exercise. The virtual intervention group will combine participants across both study locations and run sessions when sufficient numbers are recruited. Self-management education content will be unchanged to the in-person sessions but conducted over a virtual platform (i.e., videoconferencing) with participants also attending virtually.
  Interventions: Behavioral: Virtual rehabilitation group

INTERVENTIONS:
Behavioral: In-person rehabilitaiton group — participants who have chosen to complete the study intervention by coming in for their 8 week education and exercise sessions.
  Arms: In-person Intervention arm
Behavioral: Virtual rehabilitation group — Participants who have chosen to complete the study virtually instead of in-person sessions.
  Arms: Virtual Intervention arm

SUMMARY:
The proposed study is a Phase II, feasibility, randomized controlled preference based study. This will be conducted in Vancouver and Toronto and includes breast and colorectal cancers.

DETAILED DESCRIPTION:
Cancer rehabilitation interventions that address common impairments and focus on maintaining or reducing the rate of functional decline are greatly needed for the growing population of cancer survivors living with incurable or metastatic cancer. In the curative setting, the main gaps in care include lack of referral and barriers to access care; however, in the metastatic setting, high quality evidence on safety, acceptability, and efficacy is still required. In response, based on the results of a need assessments (n=50) of this population and input from palliative care experts, we recently developed the CaRE-Advanced Cancer (CaRE-AC) program. Similar to CaRE@ELLICSR, CaRE-AC is an 8-week multidimensional, group-based program with exercises classes and selfmanagement skills teaching. A single-arm phase I pilot of this program is currently being conducted to assess the feasibility and acceptability (Co-PIs Jones/Langelier). To date, 14 patients have enrolled and 9 patients have completed the program (64%). All participants reported feeling the program was safe and 90% were satisfied with the structure and content.

Data collection is expected to be complete be the end of 2019 and the findings will inform revisions to the program format and content. To build on this work, Project Three is a Phase II feasibility RCT of the CaRE-AC program. Results will inform the development of a multicentre pragmatic RCT protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosed with locally advanced incurable or metastatic breast or colorectal cancer
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Fully independent with ambulation and transfers with or without ambulatory assistance
* Palliative Performance score of >70 (moderate predictive power estimating life expectancy >6 months)
* Receiving first or second line anti-cancer treatments in the metastatic / incurable setting (a relative proxy for expected survival >6 months)
* Medical clearance to participate from treating physician

Exclusion Criteria:

* Wheelchair level community ambulation
* Moderate or severe non-cancer pain (>6 out of 10 on visual analog scale)
* Moderate or severe cancer bone pain (>Gr 2 bone pain (i.e., moderate pain limiting instrumental ALDs or worse) as measured on CTCAE (see below))
* Severe or uncontrolled depressive symptoms (>20 on PHQ-9)
* Known neurological conditions influencing cognition and preventing safe or appropriate engagement with self-management and exercise recommendations (e.g., dementia, traumatic brain injury, or brain metastasis influencing cognition or causing moderate-to-severe motor-sensory-coordination). Best determined by the referring physician or nurse practitioner.
* Unable to communicate sufficiently in English to complete intervention, questionnaires, and consent.
* Unwillingness to be randomized, participate in a group intervention, or attend individual physical assessments.
* Inability to operate videoconferencing if preference is virtual programming.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Drop-out rates as a measure of feasibility (demand/update of intervention) | 6 months
  Number of patients who complete the study/ drop-out will be used to identify feasibility of the intervention.
Patient preference as assessed during clinical support as a measure of feasibility (acceptability) | 6 months
  Check-ins with Kinesiologist during assessments will be used to identify intervention acceptability/preference.
Measuring safety/practicality as assessed during one-on-one with the health coach (analyzed as qualitative data) | 6 months
  Completed over MS Teams/in-person and will be a conversational question and answer format.

SECONDARY OUTCOMES:
Demographics | 6 months
  Demographic details will be collected from participants at the time of initial assessment via an intake questionnaire. There are no scales, only patient reported outcome questions.
Disability | 6 months
  Measured using the 12 item World Health Organization Disability Assessment Schedule 2.0 which is a cross-cultural, standardized method for measuring limitations and restrictions on individuals' activities and participation in society.
Physical functioning | 6 months
  Measured using the 10 item physical function subscale of Short-Form Health Survey (scale from 0 (negative health) to 100 (positive health) ).
Social functioning | 6 months
  Measured using the Social difficulties Inventory. A 0.0 score indicates perfect comparison with consensus group and > or equal to 2 indicates unacceptable performance/remedial action required
Depression | 6 months
  Measured using the Patient Health Questionnaire. The test is scored on a scale from 0 to 27, with higher scores indicating more severe symptoms.
Anxiety | 6 months
  Measured using the Generalized Anxiety Disorder 7. The overall GAD 7 score ranges between 0 and 21, 0 meaning no anxiety and 21 meaning severe anxiety.
Physicial activity | 6 months
  Measured using the modified Godin Leisure Score Index (LSI) of the Godin and Shepherd Leisure Time Exercise Questionnaire (GLTEQ)
Quality of Life for advanced cancer - daily life activities | 6 months
  Measured using EuroQol 5 dimension. This measure has 5 levels, with level 1 indicating no problems and level 5 indicating extreme problems
Quality of Life for advanced cancer - wellbeing | 6 months
  Measured using Functional Assessment of Chronic Illness Therapy-Palliative Care. This is a measure of health-related quality of life for persons with advanced cancer.
Symptom Burden | 6 months
  Measured with the 9-item Edmonton Symptom Assessment System. Each symptom is rated from "0 to 10". A score of "0" means you do not have the symptom. A score of "10" means that your symptom is at its very worst.
Safety and Health Care Utilization | 6 months
  Measured using a self-report questionnaire. tilization can be measured as the number of services provided to a patient, such as the number of X rays. More often, however, a variety of procedures and services are of interest, and some measure of "cost" is assigned to each service so that resource intensity can be summed over all provided services.
Weekly Session feedback | 8 weeks
  Following each educational module, participants will be asked to complete a short feedback form of 7-10 questions. Questions will explore participant's feelings surrounding session length, content, presentation quality, and recommendations for improvement. Additional questions for participants in the virtual arm will be included and inquire about video, audio, and presenter quality.
Physiological measure of height | 6 months
  Participant height at baseline
Physiological measures of weight | 6 months
  Participant weight at all physical assessments (T1, T3, T4, T5, not T2) will be collected. This data will inform calculations for BMI.
Physiological measures of exercise Intensity (Perceived Exertion) | 6 months
  During each exercise class participants will be instructed on the target rated perceived exertion (RPE) goal for that day. The RPE has been found to provide a good estimate of participant heart rate during physical activity54. Following each exercise class, each participants will be asked to provide exercise staff with a RPE score on a scale of 6 (no exertion at all) to 20 (maximal exertion) of effort. Participants who do not achieve the target RPE will be asked to provide a reason (if known).
Physiological measures of total Exercise Participation for sleep | 6 months
  Each participant will be provided a FitBit® to help track purposeful and leisure time physical activity from time point T1 (program intake) through T4 (3 months post program completion). From those consenting, data pertaining to step count sleep will be downloaded from participant accounts at each time point (T2, T3, and T4).
Physiological measures of total Exercise Participation for step count | 6 months
  Each participant will be provided a FitBit® to help track purposeful and leisure time physical activity from time point T1 (program intake) through T4 (3 months post program completion). From those consenting, data pertaining to step count will be downloaded from participant accounts at each time point (T2, T3, and T4).
Physiological measures of total Exercise Participation for heart rate. | 6 months
  Each participant will be provided a FitBit® to help track purposeful and leisure time physical activity from time point T1 (program intake) through T4 (3 months post program completion). From those consenting, data pertaining to heart rate will be downloaded from participant accounts at each time point (T2, T3, and T4).
Physiological measures of cardiorespiratory fitness | 6 months
  Measured with the six minute walk test (6MWT)
Physiological measures of muscular strength | 6 months
  Measured with hand grip strength for upper body
Physiological measures of endurance | 6 months
  Measured with 30-second sit to stand test for lower body strength
Physiological measures of balance | 6 months
  Measured with the Balance test
Physiological measures of Performance | 6 months
  Measured with the 4-meter Gait speed test

OTHER OUTCOMES:
Performance Status | 6 months
  Performance Status - Measured with the Palliative Performance Scale version 2.0. The scale ranges from 0% to 100% with zero indicating death and 100% indicating normal/no evidence of disease.
Measure of performance status | 6 months
  The Eastern Cooperative Oncology Group measure of performance status describes a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.). The scale runs from 0 to 5, with 0 denoting perfect health and 5 death.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Jones, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada